CLINICAL TRIAL: NCT05876793
Title: Effective Dose of Remiazolam Tosylate Combined With Propofol in Upper Gastrointestinal Endoscopy Sedation: a Dose-determination Study Using Dixon's Up-and-down Method
Brief Title: Effective Dose of Remimazolam Combined With Propofol in Painless Gastroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Mengchang Yang, M.D., Sichuan Provincial People's Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HR7056+propofol
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Effect of Drug
Keywords: combination; effective dose; remimazolam; propofol

STUDY DESIGN:
Intervention Model Description: We will use the Dixon's up and down method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- remimazolam tosylate (Experimental): The fixed dose of propofol in this study was 0.5mg/kg, with an injection time of 30 seconds. Subsequently, remimazolam was administered at an initial dose of 0.1mg/kg. After 1 minute of administration, sedation was evaluated using MOAA/S. When the MOAA/S score was ≤ 1, endoscopic examination could begin. If the patient did not show physical activity or coughing, sedation was considered successful, and the next patient's medication dose was reduced by 0.02mg/kg; On the contrary, if sedation fails, the next patient will receive an additional 0.02mg/kg of medication.
  Interventions: Drug: Remimazolam tosilate

INTERVENTIONS:
Drug: Remimazolam tosilate — The fixed dose of propofol in this study was 0.5mg/kg, with an injection time of 30 seconds. Subsequently, remimazolam was administered at an initial dose of 0.1mg/kg. After 1 minute of administration, sedation was evaluated using MOAA/S. When the MOAA/S score was ≤ 1, endoscopic examination could begin. If the patient did not show physical activity or coughing, sedation was considered successful, and the next patient's medication dose was reduced by 0.02mg/kg; On the contrary, if sedation fails, the next patient will receive an additional 0.02mg/kg of medication.Successful sedation results in a positive reaction, while failure results in a negative reaction. This study ends when 7 positive and negative reactions intersect

SUMMARY:
This study used sequential method（Dixon's up and douwn） to determine the effective dose of remiazolam combined with propofol in painless upper gastrointestinal endoscopy

DETAILED DESCRIPTION:
Remimazolam tosylate is a novel benzodiazepine drug that can be used for gastrointestinal sedation. However, some studies have reported that the sedative effect of using remimazolam alone is poor, and the patient's body movements are obvious, which affects the operation of endoscopists. Propofol, as a commonly used sedative drug, has good sedative effects, but has a high incidence of adverse events, especially cardiovascular system inhibition. Therefore, this study will explore the effective dose of remimazolam combined with propofol, reduce the adverse events of propofol and increase the sedative efficacy of remimazolam. This study only set up one study group, fixed the dosage of propofol, adjusted the dosage of Remimazolam to meet the appropriate sedation requirements for patients. Patients with successful sedation were judged to have a negative reaction, while patients with failed sedation were judged to have a positive reaction. A sequential chart was drawn based on the sedation situation until 7 positive negative reaction intersections were found, and the study ended

ELIGIBILITY:
Inclusion Criteria:

* ASA grading I to II, with a BMI of 18 to 30 kg/m2

Exclusion Criteria:

* Uncontrolled severe hypertension, previous history of abnormal anesthesia, unstable angina and myocardial infarction, abnormal liver and kidney function, acute upper respiratory tract infection, suspected difficulty in the airways, allergies to opioids, milk, eggs, and propofol, long-term use of sedative and analgesic drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of body movements or coughing | Day 1
  Incidence of body movements or coughing=（Number of people experiencing physical activity or coughing/total number of people studied）

SECONDARY OUTCOMES:
Sedation success time | Day 1
  MOAA/S≤1
Inspection time | Day 1
  The time from the beginning of the endoscopy to the exit of the examination mirror from the oral cavity
full alert time | Day 1
  The time from the last administration to the first MOAA/S score of 5 points when the patient reaches 5 points in three consecutive MOAA/S scores
incidence of adverse events | Day 1
  Mainly including respiratory adverse events and circulatory adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China